CLINICAL TRIAL: NCT01030757
Title: Phase II Study of Stereotactic Body Radiation Therapy Using Tomotherapy for Metastatic Tumors to the Liver
Brief Title: Study of Stereotactic Body Radiation Therapy Using Tomotherapy for Metastatic Tumors to the Liver
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0819; NCI-2011-02945 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Liver Cancer
Keywords: Liver Cancer; Metastatic Liver Cancer; Tomotherapy; Stereotactic Body Radiation Therapy
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tomotherapy (Experimental): Intervention: Stereotactic Body Radiation Therapy using Tomotherapy. Tomotherapy treatment: A total of 60 Gy using 12 Gy per fraction over 5 fractions to be given within 10 calendar days. Each fraction of 12 Gy will be divided into 2 fractions of 6 Gy given in one day within 6 hours. Dose will be prescribed to the isodose line which covers at least 90% of the PTV.
  Interventions: Radiation: Tomotherapy treatment

INTERVENTIONS:
Radiation: Tomotherapy treatment — * A total of 60 Gy using 12 Gy per fraction over 5 fractions to be given within 10 calendar days
  * Each fraction of 12 Gy will be divided into 2 fractions of 6 Gy given in one day within 6 hours
  * Dose will be prescribed to the isodose line which covers at least 90% of the PTV
  * Dose homogeneity +/- 5%

SUMMARY:
The purpose of this study is to determine the response of liver tumors to radiation therapy using Tomotherapy.

DETAILED DESCRIPTION:
The purpose of this study is to determine the response of liver tumors to radiation therapy. This study will be using a type of radiation therapy called tomotherapy. Tomotherapy is a relatively new kind of therapy which is able to focus a large amount of radiation to a small area with relatively less radiation to the surrounding non-cancerous part of the organ. This study is being done to find out if this technique is able to control the cancer better or not than the standard radiation and also to study its safety. The usual treatment for this type of disease for patients who are eligible is surgery to remove the tumors. For patients who aren't eligible for surgery or who chose not to have surgery, they are treated with low daily doses of radiation given over many weeks; however this type of treatment has not been very effective.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of solid primary tumor metastatic to liver
* Age greater than or equal to 18 years old
* Zubrod performance status less than or equal to 1
* Negative pregnancy test for women of child bearing potential
* Informed consent
* Less than or equal to 3 liver metastases
* Each lesion must be less than or equal to 6 cm in maximal diameter
* No prior radiation to lesions being treated
* Patient is not a surgical candidate or refuses surgery
* Absolute neutrophil count ≥ 1800
* Platelets ≥ 100000
* Hemoglobin ≥8.0
* Systemic therapy (chemotherapy) completed at least 2 weeks prior to SBRT
* At time of radiation treatment planning, at least 700 cc of normal liver must receive less than 15 Gy

Exclusion Criteria:

* Contraindications to radiation
* Pregnant or lactating females who chose to breast feed
* Patients must have recovered from toxicity of prior therapy
* Any co morbid condition that' in the view of the attending physician' renders the patient at high risk from treatment complications
* Patients currently receiving anticoagulation with coumadin or IV heparin
* Liver cirrhosis
* Clinical ascites
* Bilirubin > 3, Albumin < 2.5, liver enzymes 3 times above normal, Creatinine > 1.8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Liem, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States

REFERENCES:
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8 subjects were screened; 6 did not meet entry criteria. 2 subjects were enrolled
Groups:
- Tomotherapy: Intervention: Stereotactic Body Radiation Therapy using Tomotherapy. Tomotherapy treatment: A total of 60 Gy using 12 Gy per fraction over 5 fractions to be given within 10 calendar days. Each fraction of 12 Gy will be divided into 2 fractions of 6 Gy given in one day within 6 hours. Dose will be prescribed to the isodose line which covers at least 90% of the PTV.
  Tomotherapy treatment: -A total of 60 Gy using 12 Gy per fraction over 5 fractions to be given within 10 calendar days
  * Each fraction of 12 Gy will be divided into 2 fractions of 6 Gy given in one day within 6 hours
  * Dose will be prescribed to the isodose line which covers at least 90% of the PTV
  * Dose homogeneity +/- 5%
Period: Overall Study
Arm/Group | Tomotherapy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tomotherapy
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 73 [68 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate (Complete Response + Partial Response).
Time Frame: 1 year
Population: Study was terminated due to low accrual; no results to report
Arm/Group | Tomotherapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Toxicity, Progression Free Survival, Clinical Benefit Rate (Complete Response + Partial Response + Stable Disease), Median Duration of Clinical Benefit, and Median Overall Survival of Subjects.
Time Frame: 1 year
Population: Study was terminated due to low accrual; no results to report.
Arm/Group | Tomotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Tomotherapy
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes